CLINICAL TRIAL: NCT03446339
Title: Territory-Wide Pulmonary Hypertension Screening Amongst Patients With Connective Tissue Diseases: A Prospective Screening Study
Brief Title: Pulmonary Hypertension Screening for Rheumatology Patients (SOPHIE)
Acronym: PAH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Chung-Wah David SIU, Professor, The University of Hong Kong
Other Study IDs: PH_Screening_1.4.2017 ver.1
Record Dates: First submitted 2018-01-29; First posted 2018-02-26 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Connective Tissue Diseases; Systemic Sclerosis; Systemic Lupus Erythematosus
MeSH Terms: conditions — Connective Tissue Diseases; Scleroderma, Systemic; Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pulmonary arterial hypertension (PAH) is a serious and often fatal complication of connective tissue diseases including systemic sclerosis and systemic lupus erythematosus. It has been reported primarily from European series that the prevalence of PAH in patients with connective tissue diseases particularly systemic sclerosis is as high as 15-20%. However, given the paucity of medical literature in the area from Chinese population, the prevalence of PAH amongst Chinese patients with these conditions is largely unknown. Even worse, PAH is often undiagnosed amongst patients with connective tissue diseases due to the lack of awareness and/or access to echocardiography, which is a non-invasive first-line screening tool for PAH. As a result, most patients at diagnosis of PAH are at a relatively late stage, rendering pharmacological treatment less effective. Here, the investigators propose a territory-wide pulmonary hypertension screening for patients with connective tissue disease in order to (1) detect pulmonary hypertension amongst patients with connective tissue disease through systematic screening, and (2) understand the prevalence of pulmonary hypertension in Chinese patients with connective tissue diseases.

DETAILED DESCRIPTION:
Objectives:

1. To detect pulmonary hypertension amongst patients with connective tissue diseases through systematic screening
2. To understand the prevalence of pulmonary hypertension in Chinese patients with connective tissue diseases

Study design:

The study is a territory-wide pulmonary hypertension screening project. Patients fulfilling the inclusion and exclusion criteria will undergo screen echocardiography as baseline to detect subclinical pulmonary hypertension.

Screening procedure:

Participants will undergo usual clinical assessment by the rheumatology teams of the parent hospitals including standard 12-lead ECG and 6-minute hall walk distance. then they will be referred to the Division of Cardiology, the Department of Medicine, the University of Hong Kong for (1) Echocardiography and (2) BNP (or pro-NT BNP) assay. The echocardiography will be performed based on the European Society of Cardiology (ESC)/European Respiratory Society (ERS) Guidelines. The echocardiographic probability of pulmonary hypertension will be determined (low, intermediate, and high).

Statistical analysis and power calculation:

There are no studies on which to calculate a power equation, because there are no previous reports on the prevalence of pulmonary hypertension in Chinese rheumatological patients. The sample size is based on our local prevalence of the rheumatological diseases.

Continuous variables will be expressed in mean ± SD. Statistical comparisons were performed using Student's t test or Fisher's exact test, as appropriate. The outcomes would be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patientw with either (1) systemic lupus erythematosus, (2) systemic sclerosis, or (3) other connective tissue diseases at risk of pulmonary hypertension
* Voluntarily agrees to participate by providing written informed consent
* Age ≥ 18 at enrolment

Exclusion Criteria:

- Refuse to participate the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1,800 rheumatology patients with connective tissue diseases from public hospitals within Hospital Authority of Hong Kong
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2017-08-03 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of asymptomatic pulmonary hypertension in Chinese patients with connective tissue diseases | 36 months
  Proportion of patients diagnosed to have pulmonary hypertension

SECONDARY OUTCOMES:
Clinical predictor of Echocardiography for pulmonary hypertension in Chinese patients with connective tissue diseases | 36 months
  Cardiac functional and structural data for pulmonary hypertension detection
Clinical predictor of BNP assay for pulmonary hypertension in Chinese patients with connective tissue diseases | 36 months
  Cardiac marker for cardiac problems indication

CONTACTS AND LOCATIONS:
Overall Officials: David Chung-Wah Siu, Professor, Principal Investigator — The Universtiy of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, China